CLINICAL TRIAL: NCT00463528
Title: Women and Childres at the Focal Point for the Schistosomiasis Control and Sustainability and Effectiveness in the Hydro Agricultural Zone of Sourou, Burkina Faso
Brief Title: Women and Children as the Focus for Control of Schistosomiasis Infections in the Irrigations Area of Burkina Faso
Status: Completed | Type: Observational
Sponsor: DBL -Institute for Health Research and Development (Other)
Other Study IDs: SRP-BF-JNP-05
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Schistosomiasis
Keywords: schistosomiasis; gender perspectives
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of this study is to examine the extent of schistosomasis infections in women and children, their daily activites that encumber contact with water and their knowledge and attitudes towards the prevention of schistosomiasis.

The hypothesis that will be explored is that women and children spent more time with agricultural and household activities which bring them in contact with water and therefore give them an increased risk of being infected by schistosoma. Prevention and control of schistosomiasis has to be focusing on women and children.

DETAILED DESCRIPTION:
The study will be carried out in and irrigation area of Burkina Faso where people relay on water. The study applies several methodes;

1. Parasitological survey: From thre villages 200 women and children are randomly sampled to have their urin and stool examined for parasittes.
2. Observations: At each village sites at the irrigation canals where people meet and have their activities observations of the kind and the duration of watercontact will be observed.
3. Focus group interview: In each village 5 focus group interviews will be conducted with 6 to 12 participants in each group
4. Individual interviews: for the participant in the focus group interview a total of 45 participants will be selected for indept individual interviews
5. Questionnaire: a total of 360 questionnairs will be distributed to participants in the parasitological survey, the focus group interviews and to participants who did not participate in any of the above mentioned.

Participants will be women and children from the three villages.

ELIGIBILITY:
Inclusion Criteria:

Women and children from three villages

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-12; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean N Poda, Ph.d.,M.Sc., Principal Investigator — Institute of Health Sciences Research, Burkina Faso